CLINICAL TRIAL: NCT00665743
Title: An Open-Label, Randomized, 3-Way Crossover Study to Evaluate the Relative Bioavailability of a Single Oral Dose of Naproxen 500 mg Administered as PN 400 (Naproxen / Esomeprazole), as the [Active Comparator 1], or as [Active Comparator 2] in Healthy Volunteers
Brief Title: Study Evaluating the Bioavailability of Naproxen 500 mg in Three Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: David Taylor, Pozen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PN400-102
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): PN400 (naproxen/esomeprazole)
  Interventions: Drug: PN400
- B (Active Comparator): naproxen 500 mg
  Interventions: Drug: naproxen
- C (Active Comparator): naproxen 500 mg
  Interventions: Drug: naproxen

INTERVENTIONS:
Drug: PN400 — naproxen 500 mg /esomeprazole 20 mg
  Arms: A
Drug: naproxen — naproxen 500 mg tablet
  Arms: B
Drug: naproxen — naproxen 500 mg
  Arms: C

SUMMARY:
We will evaluate the bioavailability of naproxen 500 mg administered as three dfferent formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects between 18-55 years of age as well as other standard inclusion criteria for a study of this nature

Exclusion Criteria:

* Standard exclusion criteria for a study of this nature

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess and compare the pharmacokinetics and relative bioavailability of a single oral dose of naproxen 500 mg administered in 3 formulations | 72-hour PK

SECONDARY OUTCOMES:
To evaluate the safety of the 3 treatments | entire study duration

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States